CLINICAL TRIAL: NCT05386225
Title: Individualized Follow-Up for Head and Neck Cancer
Acronym: INFLUENCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Betaalbaar Beter (VGZ) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 112491
Record Dates: First submitted 2022-05-06; First posted 2022-05-23 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancer
Keywords: Follow-Up Care; Follow-Up Studies
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standardized follow-up: Participants who chose to continue guideline-prescribed, standardized follow-up one year after HNC treatment.
- Individualized follow-up: Participants who chose to switch to individualized follow-up one year after HNC treatment. Follow-up visits will only be scheduled based on clinical symptoms and questions, initiated by the patient.

SUMMARY:
This pilot study evaluates offering Head and Neck Cancer (HNC) patients a choice between standardized and individualized follow-up after HNC treatment. Following treatment, the patient will be educated about self-examination of the head and neck and which physical symptoms require a follow-up visit. After completing 1.5 years of uncomplicated guideline-prescribed follow-up, patients will be offered the option to switch to individualized follow-up through a tailored decision aid. Standardized follow-up entails continuing the guideline-prescribed follow-up schedule until five years after treatment. Individualized follow-up consists of follow-up visits based on symptoms and other needs at the patient's initiative. We hypothesize that giving patients the choice between standardized and individualized follow-up is feasible and saves costs while maintaining quality of life.

DETAILED DESCRIPTION:
Background of the study:

Head and Neck Cancer (HNC) patients are currently enrolled in routine follow-up by medical specialists (standardized follow-up) for five years after primary treatment, according to the Dutch guideline Head and Neck Tumors. Similar recommendations are described in guidelines from the US and UK. The purposes for aftercare following cancer treatment as stated by the Health Council of the Netherlands are to address the effects of the disease and treatment itself, to detect new cancer manifestations, and to evaluate medical procedures to improve the quality of care.

The majority of HNC recurrences occur in the first 1.5-two years after treatment, and most of them cause clinical symptoms.It has not been proven that patients with recurrent disease discovered in the asymptomatic phase have better treatment options and life expectancy than patients who experience symptoms at the time of discovery.

Detecting second primary tumors (SPT) is an extra argument for routine follow-up as HNC patients are at greater risk of developing second primary cancers. SPTs are known to negatively affect overall long-term survival, especially those found outside the head and neck area. However, the way in which control visits are performed, namely physical examination of the head and neck, does not aim to identify SPTs elsewhere in the body. Because the incidence of SPTs remains stable over the years after treatment, detecting them would require life-long follow-up through diagnostic imaging.

Many patients express the concern that their cancer will progress or recur after treatment, also known as fear of cancer recurrence (FCR). FCR has a major impact on quality of life. It is not clear whether routine control visits exacerbate or relieve FCR, although previous research suggests that patient-led follow-up, in which prescheduled visits are replaced by patient-education and access to care by self-referral, does not influence FCR. Furthermore, patients have reported being anxious before scheduled control visits.

Overall, de-intensifying routine follow-up after primary HNC treatment seems to be sensible in the light of discovering recurrent or new cancers and will probably not affect FCR. However, reducing the frequency of prescheduled control visits for all HNC patients may deny the varying needs of individual patients. These needs include receiving more information about the treatment trajectory and being more involved in the decision-making process. Therefore, we have implemented a novel decision-aided follow-up program that allows HNC patients to choose between continuing standardized follow-up with prescheduled control visits, and individualized follow-up with symptom-based visits.

Objective of the study:

The aim of this project is to evaluate implementing the choice for individualized follow-up after head and neck cancer treatment at the Radboudumc and Rijnstate, the preferred partner of the Radboudumc regarding head and neck oncology. It will be investigated to what extent it is feasible to offer patients the choice for individualized follow-up, 1.5 years after completion of treatment. In addition, insight into (cost-)effectiveness is explored.

Primary research question: What is the feasibility of offering head and neck cancer patients the choice between standardized and individualized follow-up in a shared-decision making process supported by a decision-aid after completing 1.5 years of standardized follow-up?

Secondary research questions:

1. How many patients choose individualized follow-up after completing 1.5 years of standardized follow-up if they are supported by a decision-aid and their treating physician in a shared-decision-making process?
2. To what extent do patients who choose individualized follow-up differ from patients who choose standardized follow-up, based on gender, age, educational level, or other patient- or tumor characteristics?
3. What are patients' experiences with the choice in terms of the decision-making-process and decisional regret?
4. What are physicians' experiences with the choice in terms of the decision-making-process?
5. What is the effect of this choice on fear of cancer recurrence and other quality of life outcome measures?
6. What is the difference in costs between standardized and individualized follow-up?
7. Is there a difference in timing and manner of detection of recurrences between patients who opted for standardized and individualized follow-up? We hypothesize that giving patients the choice between standardized and individualized follow-up is feasible and has a positive effect on FCR, while maintaining QoL and reducing medical costs. We do not expect to diagnose less recurrences or second primary tumors in patients who opted for individualized follow-up.

Study design:

This is an observational study (prospective cohort study) to evaluate offering a choice for individualized follow-up after treatment for HNC in Radboudumc and Rijnstate.

Study population:

Patients with a primary malignancy in the head and neck region (nose, nasopharynx, nasopharynx, oral cavity, pharynx, larynx) who have undergone treatment with curative intent.

Introducing individualized follow-up:

All head and neck cancer patients who are enrolled in standardized follow-up will be informed on the choice between standardized and individualized follow-up directly after treatment. Patients who have completed 1.5 years of standardized follow-up will be asked to make a choice between continuing standardized follow-up or switching to individualized follow-up. Patients will gain access to our online decision-aid to support the decision-making process. Their treating physician will explain all the details during a decision-making consult, after which a decision is made.

Including participants:

Patients who are eligible to participate in this study will be scheduled for an outpatient visit with an independent researcher 1.5 years after treatment, regardless of their choice for standardized or individualized follow-up. The researcher will explain the study and study-goals. Another appointment will be scheduled two weeks later to answer possible questions and, if the patient is willing to participate, obtain informed consent.

Ethical aspects:

We expect that patients who are given the opportunity to choose their own form of follow-up will not regret their decision. Nevertheless, participants always have the option to withdraw their decision at any time during the study, and afterwards. Participants in this study will not receive any special compensation or reward.

Data management:

All participants who have given informed consent are assigned an identification code. The identification code is copied on the code list. Identifiable data of the included study participants are kept in the code list (name, address, telephone number, medical file number (MDN), etc.). No traceable data are recorded in the electronic database (Castor EDC), only the participant's identification code. The code list is kept in a separate and secured digital environment.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor of the head and neck
* First primary HNC
* Participant was treated with curative intent
* Participant has completed one year of uncomplicated routine follow-up
* Treating physician supports the possible choice for patient-led follow-up

Exclusion Criteria:

* Malignant tumors of salivary glands
* Participant is cognitively impaired
* Participant is unable to read or write in Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the Radboud University Medical Center, which is one of eight specialized head and neck oncology care centers in the Netherlands, and their preferred partner Rijnstate Ziekenhuis in Arnhem, The Netherlands.
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Follow-up decision | Baseline
  The type of follow-up that was chosen (standardized or individualized) will be distracted from the electronical patient record.
Demand - assessed by the reach | 1.5 years
  Number of patients who received the decision-aid and the choice for follow-up in our clinical practice divided by the number of patients eligible to use the decision-aid and thus make a choice between the two follow-up programs.
Acceptability - assessed by the SUS | Baseline
  The use of the decision-aid will be evaluated using the System Usability Scale (SUS): 10 items giving a global view of subjective assessments of usability of the decision-aid on a 5-point scale from strongly disagree (1) to strongly agree (5). A higher score means higher usability. 10 self-constructed questions about the presentation, actual use, and perceived added value are added to the questionnaire.
Tailored decision aid - usability | Baseline
  The use of a tailored decision aid to support the decision making process will be evaluated using the System Usability Scale (SUS): 10 items giving a global view of subjective assessments of usability of the decision-aid on a 5-point scale from strongly disagree (1) to strongly agree (5).
Tailored decision aid - use and added value | Baseline
  The use of a tailored decision aid to support the decision making process will be evaluated by a self-constructed questionnaire consisting of 10 additional questions about the presentation, actual use, and the perceived added value of the decision aid from a patient perspective. A higher score means higher usability.
Tailored decision aid - implementation in clinical practice | 1.5 years
  The use of a tailored decision aid from a physician perspective will be evaluated by an adjusted version of the MIDI questionnaire to measure determinants associated with successful implementation of the decision aid. In general, a higher score means higher (expected) use in clinical practice.

SECONDARY OUTCOMES:
Quality of life - Fear of cancer recurrence | Baseline
  Fear of cancer recurrence is measured using the Cancer Worry Scale (CWS): 6 items on worries after cancer treatment rated on a 4-point scale from almost never/not at all (1) to almost always/very much (4). A high score means higher FCR.
Quality of life - EORTC QLQ C-30 | Baseline
  Quality of life is measured using the European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ C-30): 30 items organized in 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (pain, fatigue, emesis), and a global health and QoL scale rated on a scale from 0 to 100 (100 meaning perfect quality of life for functional scales or heavy burden for symptom scales).
Quality of life - EORTC QLQ-H&N35 | Baseline
  Quality of life is measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire module for patients with head and neck cancer (EORTC QLQ-H&N35): 7 multi-item scales (pain, swallowing, senses, speech, social eating, social contact, sexuality) and 11 single items (teeth, mouth opening, dry mouth, sticky saliva, coughing, feeling ill, use of pain killers, nutritional supplements, feeding tube, weight loss and weight gain) rated on a scale from 0 to 100.
Quality of life - EQ-5D-5L | Baseline
  Quality of life is measured using the EuroQuality of Life Five Dimensions (EQ-5D-5L) questionnaire, consisting of descriptive health status and visual health status. Descriptive health status: 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) rated from 1 (no problems) to 5 (extreme problems).
  Visual health status: visual analogue scale (VAS) from 'worst health you can imagine' - 'best health you can imagine'.
Quality of life - Fear of cancer recurrence | 1.5 years
  Fear of cancer recurrence is measured using the Cancer Worry Scale (CWS): 6 items on worries after cancer treatment rated on a 4-point scale from almost never/not at all (1) to almost always/very much (4). A high score means higher FCR.
Quality of life - QLQ C-30 | 1.5 years
  Quality of life is measured using the European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ C-30): 30 items organized in 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (pain, fatigue, emesis), and a global health and QoL scale rated on a scale from 0 to 100 (100 meaning perfect quality of life for functional scales or heavy burden for symptom scales).
Quality of life - QLQ-H&N35 | 1.5 years
  Quality of life is measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire module for patients with head and neck cancer (EORTC QLQ-H&N35): 7 multi-item scales (pain, swallowing, senses, speech, social eating, social contact, sexuality) and 11 single items (teeth, mouth opening, dry mouth, sticky saliva, coughing, feeling ill, use of pain killers, nutritional supplements, feeding tube, weight loss and weight gain) rated on a scale from 0 to 100.
Quality of life - EQ-5D-5L | 1.5 years
  Quality of life is measured using the EuroQuality of Life Five Dimensions (EQ-5D-5L) questionnaire, consisting of descriptive health status and visual health status. Descriptive health status: 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) rated from 1 (no problems) to 5 (extreme problems).
  Visual health status: visual analogue scale (VAS) from 'worst health you can imagine' - 'best health you can imagine'.
Shared decision making for patients | Baseline (after decision making consult)
  Shared decision making will be evaluated using the Shared Decision Making Questionnaire (SDM-Q-9) for patients: 9 items on SDM rated on a 6-point scale from completely disagree (0) to completely agree (6) from a patient perspective.
Shared decision making for physicians | Baseline (after decision making consult)
  Shared decision making (routine or patient-led follow-up) will be evaluated using the Shared Decision Making Questionnaire (SDM-Q-9) for physicians: 9 items on SDM rated on a 6-point scale from completely disagree (0) to completely agree (6) from a physician perspective.
Decisional conflict | Baseline
  Decisional conflict is measured by the Decisional Conflict Scale (DCS): 16 items considering decisional conflict rated on a 5-point scale from strongly agree (0) to strongly disagree (4). A high score means higher decisional conflict.
Decisional regret | 1.5 years
  Decisional regret is measured by the Decisional Regret Scale (DRS): 5 items considering decisional regret rated on a 5-point scale from strongly agree (0) to strongly disagree (4). A high score means higher decisional regret.
Practicality - Medical consumption | Baseline
  Medical consumption will be measured using the iMedical Consumption Questionnaire (iMCQ): 31 items to assess patient reported general medical consumption (primary and secondary care, including medicine use).
Practicality Medical consumption | 1.5 years
  Medical consumption will be measured using the iMedical Consumption Questionnaire (iMCQ): 31 items to assess patient reported general medical consumption (primary and secondary care, including medicine use).
Practicality - Productivity loss | Baseline
  Productivity loss will be measured using the iProductivity Cost Questionnaire (iMCQ): 18 items to assess patient reported productivity losses in hours (considering absenteeism, presenteeism, and unpaid work).
Practicality - Productivity loss | 1.5 years
  Productivity loss will be measured using the iProductivity Cost Questionnaire (iMCQ): 18 items to assess patient reported productivity losses in hours (considering absenteeism, presenteeism, and unpaid work).
Practicality - outpatients visits and tests | 1.5 years
  The number of outpatient visits and diagnostic tests during the follow-up year after the choice for individualized or standardized follow-up will be collected from the electronical patient record.

OTHER OUTCOMES:
Sociodemographic and basic clinical characteristics - input variables | Baseline
  Patient records: date of birth, sex, primary treatment hospital, date of diagnosis, clinical and pathological tumor characteristics, date and type of primary treatment.
  Patient reported: living situation, educational level, employment, smoking, alcohol consumption.
Oncological outcomes | 1.5 years
  In case of recurrent/second primary tumor(s) during the study period, the following will be retrieved from the patient record: date of diagnosis, clinical and pathological characteristics, date and type of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Takes, Prof, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available after publication of the manuscript describing the results of this study. The exact date and duration of data availability have not been established yet.
Access Criteria: Criteria for access have to be discussed by the authors.

REFERENCES:
- [Derived] van de Weerd C, van Tol-Geerdink JJ, van den Broek GB, Kaanders JHAM, Marres HAM, Hermens RPMG, Takes RP. Individualised follow-up for head and neck cancer-design of a prospective cohort study to assess its feasibility. BMJ Open. 2022 Dec 29;12(12):e068750. doi: 10.1136/bmjopen-2022-068750. PMID 36581428